CLINICAL TRIAL: NCT04405609
Title: Usability Study of "ArmAssist 2.0." Robot: Homecare Arm Rehabilitation in Acute, Subacute and Chronic Stroke Patients
Brief Title: Usability Study of "ArmAssist 2.0." Robot: Homecare Arm Rehabilitation in Stroke Patients
Acronym: PUAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: TECNALIA Research & Innovation (Unknown); GMV Innovating Solutions (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ArmAssist 2.0
Record Dates: First submitted 2020-05-19; First posted 2020-05-28 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Stroke; Rehabilitation; Upper Limb Rehabilitation; Telerehabilitation; Robot-assisted Therapy
Keywords: Stroke; Cerebrovascular Disorders; Robotic
MeSH Terms: conditions — Stroke; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ArmAssist group (Experimental): The post-stroke patients who participate in the study, are classified in differents stages (3 patients in each stage).
  Group 1: subacute, between 2 - 6 months Group 2: chronic of short evolution, between 6 - 12 months Group 3: long-term chronic, more than 12 months.
  The system is tested in a clinical (training) and patients' home setting. The ArmAssist system includes the ArmAsist 2.0 device (without motors), the tele rehabilitation platform based on serious games and Antari's HomeCare tele-care platform for the clinicians.
  Interventions: Device: ArmAssist

INTERVENTIONS:
Device: ArmAssist — The usability study protocol include 3 ArmAssist systems (2 designed for the left hand and one for the right hand) that could not be used in parallel because the aim of the study was to bring the systems to the home environment during part of the evaluation.
  The usability study is carried out in two phases:
  1. First phase: 5 weeks.
  2. Second phase: 3 weeks. Each phase included a week of training at the Hospital or IMIBIC facilities with a physiotherapist, and then 2 weeks at the patient's home, being the first one with the physiotherapist supervision and the second one by their own with the possibility of physiotherapist remote support.

SUMMARY:
The purpose of this study is to validate the usability of ArmAssist medical device, a robotic system for the rehabilitation of upper limbs in stroke patients (based on serious games). This study evaluate the usability of the system in a home environment, taking into account the ease-to-use, consistency and others; and will pretend demonstrate the feasibility of including or no, robotic therapy in home like complement of daily rehabilitation program. Finally this study investigate the acceptance from patients and therapists.

ELIGIBILITY:
Inclusion Criteria:

* Subjects over 18,
* Upper limb hemiparesis after stroke,
* Unilateral paresis and cognitive ability to understand,
* Accept and actively participate in the usability study.

Exclusion Criteria:

* Bilateral motor deficit,
* Severe spasticity,
* Psychiatric illness,
* and/or cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Quebec User Evaluation of Satisfaction with assistive Technology: QUEST scale | Through study completion, an average of 3 weeks
  The purpose of this scale is to evaluate how satisfied the patient are with the assistive device and the related services they experienced. It consists of twelve questions, eight related to the device and four related to services of 12 satisfaction items with answers from 1 'Not satisfied at all' to 5 'Very satisfied'
System Usability Scale: SUS | Through study completion, an average of 3 weeks
  This scale provides a quick, reliable tool for measuring the usability. It consists of 10 item questionnaire and answers from 1 'strongly agree' to 5 'strongly disagree'. Scores are ranging to 0-100 %, where a high score means better usability with a higher score meaning better usability
Intrinsic Motivation Inventory: IMI | Through study completion, an average of 3 weeks
  This scale is a multidimensional scale intended to assess participants subjective experience with the device (interest/enjoyment, perceived competence, effort, value/usefulness, felt pressure and tension, and perceived choice while performing a given activity). Consist of 20 item questionnaire with answers from 1 'strongly agree' to 7 'strongly disagree'.
Usability questionnaire specifically designed for the use of ArmAssist 2.0 | Through study completion, an average of 3 weeks
  It consists of a 19 item questionnaire with seven response options (Likert sacle) for respondents; from Strongly agree to Strongly disagree. To evaluate the satisfaction of patients and therapist with the system and the therapy.
Structured interviews: Willingness-to-pay questionnaire | Through study completion, an average of 3 weeks
  This interview consists in two short questions to ask to participants about the willingness-to-pay for ArmAssist 2.0. system as therapy.

SECONDARY OUTCOMES:
Fugl-Meyer Assessment (FMA) scale | Baseline, 3 weeks
  It is an index to assess the sensorimotor impairment in individuals who have had stroke. The Fugl-Meyer Assessment scale is an ordinal scale that has 3 points for each item. A zero score is given for the item if the subject cannot do the task. A score of 1 is given when the task is performed partially and a score of 2 is given when the task is performed fully. The maximun score is 66 points
Modified Asworth Scale (MAS) | Baseline, 3 weeks
  This scale measures resistance during passive soft-tissue stretching and is used as a simple measure of spasticity. It is single-item measures ranging from 0 to 4, where 0 indicates no increase in muscle tone and 4 indicates that the affected part is rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Jesus Mayordomo Riera, MD, Principal Investigator — Hospital Universitario Reina Sofia de Córdoba
Locations (1):
- Hospital Universitario Reina Sofía de Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Yes
All the collected information will be available for other researchers upon request.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Up to 12 months after trials publication.
Access Criteria: Request by e-mail to uicec@imibic.org

REFERENCES:
- [Derived] Guillen-Climent S, Garzo A, Munoz-Alcaraz MN, Casado-Adam P, Arcas-Ruiz-Ruano J, Mejias-Ruiz M, Mayordomo-Riera FJ. A usability study in patients with stroke using MERLIN, a robotic system based on serious games for upper limb rehabilitation in the home setting. J Neuroeng Rehabil. 2021 Feb 23;18(1):41. doi: 10.1186/s12984-021-00837-z. PMID 33622344